CLINICAL TRIAL: NCT01093781
Title: A Pilot Study to Evaluate the Antiproteinuric Effect of Renin Inhibition With Aliskiren in Patients With Idiopathic Membranous Nephropathy
Brief Title: Aliskiren in Patients With Idiopathic Membranous Nephropathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacturer asked to close study due to AEs experienced by subjects in other studies.
Sponsor: Mayo Clinic (Other)
Responsible Party: Fernando Fervenza, MD, PhD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-007837
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Idiopathic Membranous Nephropathy
Keywords: membranous nephropathy aliskiren proteinuria, glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, Membranous; Glomerulonephritis | interventions — aliskiren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aliskiren (Experimental): Aliskiren dose will begin with 150mg per day and later up-titrated to the maximum available dose of 300mg per day.
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren — Aliskiren dose will begin with 150mg per day and later up-titrated to the maximum available dose of 300mg per day.
  Other Names: Tekturna

SUMMARY:
The goal of this proposal is to conduct a pilot study to access the antiproteinuric effect of aliskiren in patients with idiopathic membranous nephropathy. Patients will be treated for 3 months with aliskiren aiming to achieve the maximum tolerated dose and blood pressure (>100 but <125 mmHg systolic BP >75% of the readings).

DETAILED DESCRIPTION:
In patients with nephrotic syndrome, including patients with membranous nephropathy (MN), conservative therapy consists of restricting dietary protein intake, and controlling blood pressure (target blood pressure is ≤ 125/75 mmHg), hyperlipidemia, and edema. Angiotensin-converting enzyme inhibitors (ACEi) and/or angiotensin II receptor blockers (ARB) are effective anti-hypertensive agents that can reduce proteinuria and slow progression of renal disease in both diabetic and nondiabetic chronic nephropathy patients and for these reasons they are the preferred agents to treat hypertension in proteinuric renal diseases.

Recent studies suggest that renin inhibition with aliskiren may be renoprotective and reduce proteinuria in patients with type 2 diabetes. Similar observations have also been reported in patients with membranous nephropathy and proteinuria in the range of 1-3 g/24h. These observations suggest that aliskiren may have powerful antiproteinuric. However, it is important to emphasize, that none of the patients in these studies had proteinuria greater than 3.0 g/24h. Thus, the antiproteinuric effect of aliskiren in patients with heavy proteinuria (e.g. >4g/24h) is unknown.

ELIGIBILITY:
Inclusion Criteria

* Idiopathic MN proven by diagnostic kidney biopsy.
* Age ≥18 years but ≤ 80 years.
* Proteinuria as measured by urinary protein/urinary creatinine > 4.0 on a spot sample aliquot from a 24-hour urine collection.
* Estimated GFR ≥ 30 ml/min/1.73m^2 using the 4 variable Modification of Diet in Renal Disease (MDRD) equation.

Exclusion Criteria

* Age <18 years.
* Estimated Glomerular Filtration Rate (GFR) < 30 ml/min/1.73m^2, or serum creatinine >3.0 mg/dl.
* Patient must be off prednisone, calcineurin inhibitor or mycophenolate mofetil for > 1 month and alkylating agents for > 6 months.
* Patients with presence of active infection or a secondary cause of MN (e.g. hepatitis B, HIV, systemic lupus erythematosus (SLE), medications, malignancies).
* Type 1 or 2 diabetes mellitus. Patients who have recent history of steroid induced diabetes but no evidence of diabetic nephropathy on renal biopsy performed within 6 months of entry into the study are eligible for enrollment.
* Pregnancy or nursing for safety reasons.
* Acute renal vein thrombosis documented prior to entry by renal US or CT scan.
* Previous therapy with Aliskiren

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Urine protein excretion | one year
  Urine protein excretion at 12 weeks of renin inhibition with aliskiren

SECONDARY OUTCOMES:
Blood pressure control; tolerability and side effects | one year

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Fervenza, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States